CLINICAL TRIAL: NCT06801613
Title: Correlation Between Upper Cross Syndrome and Neck Proprioception
Brief Title: Upper Cross Syndrome and Neck Proprioception
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omnia Mohamed Said El-Sayed, general practitioner, Cairo University
Other Study IDs: P.T.REC/012/005030
Record Dates: First submitted 2025-01-25; First posted 2025-01-30 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Upper Cross Syndrome
Keywords: proprioception; upper cross syndrome; neck
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- control group: Participants with UCS who do not receive the intervention (e.g., may receive standard care, education, or no treatment).
  Interventions: Other: Intervention Group

INTERVENTIONS:
Other: Intervention Group — Group/Cohort Description: Participants with Upper Cross Syndrome (UCS) who undergo the prescribed exercise or treatment protocol.

SUMMARY:
Correlation Between Upper Cross Syndrome and Neck Proprioception

Hypothesis:

No statistically significant relationship exists between upper cross syndrome and neck proprioception.

Study Design:

Randomized Controlled Trial

Participants:

Office workers (≥4h computer use/day) Age: 28-48 years Chronic nonspecific neck pain (>3 months) Forward head posture (FHP) <46° VAS score: 3-8 cm No cognitive impairments affecting participation

Exclusion Criteria:

Systemic, rheumatic, or neuromuscular diseases Neurological signs, spinal surgery, or recent physical therapy Missing ≥3 consecutive or 4 nonconsecutive sessions

DETAILED DESCRIPTION:
Study Title:Correlation Between Upper Cross Syndrome and Neck Proprioception

Hypothesis:There will be no statistically significant relationship between upper cross syndrome and neck proprioception.

Methodology:

Study Design:Randomized controlled trial

Inclusion Criteria:

Office workers using a computer for at least 4 hours daily

Aged between 28 and 48 years

Neck pain (NP) between 3 and 8 cm on a visual analog scale (VAS) (0 = no pain, 10 = unbearable pain)

Chronic nonspecific neck pain lasting for more than 3 months

Forward head posture (FHP) less than 46°

Patients willing and able to participate in an exercise program safely without cognitive impairments that would limit participation

Exclusion Criteria:

Specific causes of NP (e.g., systemic, rheumatic, neuromuscular diseases)

Central or peripheral neurological signs

Cognitive impairment

History of spinal surgery

Physical therapy treatments in the last 6 months prior to baseline assessment

Participants missing at least three consecutive or four nonconsecutive sessions

Outcome Measures:

Spinal Curvature Assessment Using Spinal Mouse DeviceThe spinal mouse device is physically guided along the skin of the spine

Neck Pain MeasurementNP is evaluated using a 10-cm VAS, a widely used clinical tool for assessing pain treatment effectiveness.

Neck Disability Index (NDI)Disability is assessed using the NDI questionnaire.

Measurement of Cervical Range of Motion (CROM) Using a CROM

Assessment of Cervical Proprioception Using the CROM DeviceHead Reposition Accuracy Tests:

Neutral Head Position (NHP) Test: Measures the ability to actively reposition the head to the self-selected neutral position.

Target Head Position (THP) Test: Measures the ability to actively reposition the head to a previously demonstrated target position.

ELIGIBILITY:
Inclusion Criteria:

* office workers (using a computer at least 4 h),

  * aged between 28 and 48 years,
  * NP between 3 and 8 cm on a visual analog scale (VAS) (from 0 indicating no pain at all to 10 indicating unbearable pain),
  * chronic nonspecific neck pain lasting for more than 3 months, and FHP less than 46° (Fathollahnejad et al., 2019).
  * Patients willing and able to participate in an exercise program safely and without cognitive impairments that would limit their participation.

Exclusion Criteria:

* specific causes of NP (e.g., systemic, rheumatic, neuromuscular diseases), central or peripheral neurological signs, cognitive impairment, spinal surgery, or physical therapy treatments in the last 6 months prior to the baseline assessment.
* Participants would be also excluded if they missed at least three consecutive or four nonconsecutive sessions (Fathollahnejad et al., 2019).

Ages: 28 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of adult office workers with specific characteristics related to their occupation, posture, and neck pain history. Below is a detailed breakdown:
  Demographic Characteristics
  Age Range: 28-48 years. Gender: Not specified, but likely includes both males and females. Occupation: Office workers using computers for at least 4 hours daily.
  Clinical Characteristics
  Chronic Nonspecific Neck Pain (CNP):
  Pain lasting ≥3 months. Pain intensity between 3-8 cm on the Visual Analog Scale (VAS).
  Forward Head Posture (FHP):
  Measured angle of FHP is less than 46°.
  No Specific Diagnoses:
  Participants with neck pain due to systemic, rheumatic, or neuromuscular diseases are excluded.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
Cervical Proprioception: | 8 weeks
  Measurement Tool: CROM device.
  Tests:
  Neutral Head Position (NHP): Assesses participants' ability to actively reposition their head to a self-selected neutral position.
  Target Head Position (THP): Assesses ability to reposition the head to a previously demonstrated target position.

SECONDARY OUTCOMES:
Neck Pain | 8 weeks
  Measurement Tool: Visual Analog Scale (10-cm scale)
  Purpose: Evaluate participants' subjective pain levels before and after the intervention.
  Scale Range: 0 (no pain) to 10 (unbearable pain). Interpretation: Higher scores indicate worse pain levels.
Balance | 8 weeks
  Measurement Tool: Biodex Balance System.
  Parameters:
  Static and dynamic balance. Postural stability score (lower scores indicate better balance). Purpose: Explore the effect of UCS on overall balance and stability.
Neck Disability Index (NDI): | 8 weeks
  Measurement Tool: NDI questionnaire. Purpose: Assess the impact of neck pain on daily activities and functional limitations.
Cervical Range of Motion (CROM) | 8 weeks
  Measurement Tool: CROM device. Purpose: Measure the range of motion in the cervical spine to detect restrictions due to UCS.

OTHER OUTCOMES:
Spinal Curvature: | 8 weeks
  Measurement Tool: Spinal Mouse Device.
  Parameters:
  Sagittal plane alignment in neutral, flexion, and extension.
  Purpose: Assess structural changes or adaptations in the spine due to UCS.